CLINICAL TRIAL: NCT06208631
Title: Effects of Haptic Movement Retraining on Osteoarthritis Progression
Brief Title: Effects of Movement Retraining on Knee Loading in Individuals With Knee Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Scott Delp, Professor of Bioengineering and Mechanical Engineering, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 34928
Record Dates: First submitted 2023-12-18; First posted 2024-01-17 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Gait modification (Experimental): Participants will learn to change muscle coordination while walking through real-time haptic biofeedback based on the activation of the gastrocnemius muscle
  Interventions: Behavioral: Gait retraining

INTERVENTIONS:
Behavioral: Gait retraining — Changing muscle coordination while walking

SUMMARY:
This study investigates how well individuals with knee osteoarthritis can learn to alter their calf muscle activation using haptic biofeedback while walking and evaluates how these changes affect knee loading.

Prior research has utilized musculoskeletal simulations to determine that reducing the activation of one of the calf muscles, the gastrocnemius, can have a large impact on reducing knee loading. However, this has not been tested in individuals with knee osteoarthritis. In this study, participants will be trained to alter the activation of their gastrocnemius muscle, by receiving haptic feedback after each step. The feedback will indicate how the participant changed their muscle activation relative to baseline. Some participants will train on a treadmill in the laboratory for up to two sessions, with 30 minutes of walking with feedback in each session. If a participant can learn to adjust their muscle activation in the first training session, they will be able to complete the second training session. Other participants will train outside the laboratory for one session with 30 minutes of walking with feedback to investigate changes in knee loading while using the new walking strategy during over-ground walking.

The movement data collected during the training sessions will be used as inputs to computer simulations of the musculoskeletal system to determine if walking with the new muscle activation strategy reduces knee loading.

ELIGIBILITY:
Inclusion Criteria:

* Medial and/or lateral compartment knee osteoarthritis
* Diagnosed with knee osteoarthritis of at least six months duration
* Ambulatory without aids
* Able to walk for at least 60 minutes
* Typical pain rating less than or equal to 4 on scale of 0-10
* Able to reduce gastrocnemius muscle activation by 10% from baseline

Exclusion Criteria:

* History of symptomatic arthritis in lower limb joints other than the knees
* Replacement of any lower extremity joint
* Symptoms originating from the patellofemoral joint
* Body mass index equal to or greater than 35
* Nerve or muscle disease associated with walking difficulty
* History of rheumatoid arthritis, gout, or autoimmune disease
* History of lower limb fracture or surgery requiring hospitalization
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2024-01-18 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in knee contact force | Evaluated during the 30 minutes of feedback walking in the second in-lab session and out-of-lab session
  Knee contact force will be evaluated using motion capture data and musculoskeletal modeling and simulations, for participants that are able to reduce gastrocnemius activation.

SECONDARY OUTCOMES:
Change from baseline in gastrocnemius activation | Evaluated during the 30 minutes of feedback walking in the first in-lab session, the second in-lab session, and the out-of-lab session
  Gastrocnemius activation measured through EMG signals.
Proportion of participants that reduce gastrocnemius activation | Evaluated during the 30 minutes of feedback walking in the first in-lab session, the second in-lab session, and the out-of-lab session
  Gastrocnemius activation will be measured through electromyography (EMG) signals, and the muscle activation during gait retraining will be compared to baseline walking. Participants that can reduce gastrocnemius activation 10% or more from baseline within 30 minutes of gait retraining will be counted as participants that can reduce gastrocnemius activation out of the total number of participants who try the gait retraining.
Proportion of participants that reduce knee contact force | Evaluated during the 30 minutes of feedback walking in the second in-lab session and the out-of-lab session
  For the participants who can successfully reduce gastrocnemius activation from baseline, knee contact force will be calculated using motion capture data and musculoskeletal modeling and simulations. The proportion of participants that reduce knee contact force from baseline during gait retraining out of the total participants that reduce gastrocnemius activation will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Scott L Delp, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford Human Performance Lab, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified experimental data and simulation results will be made available.
Time Frame: After publication and no end date
Access Criteria: Data will be publicly available online at SimTK.

REFERENCES:
- [Background] Lee KJ, Hahm KB, Kim YS, Kim JH, Cho SW, Jie H, Park CH, Yim H. The usefulness of Tc-99m HMPAO labeled WBC SPECT in eosinophilic gastroenteritis. Clin Nucl Med. 1997 Aug;22(8):536-41. doi: 10.1097/00003072-199708000-00005. PMID 9262899
- [Background] Kather L, Smidt D. [Composition of porcine uterine secretion]. Berl Munch Tierarztl Wochenschr. 1974 Oct 1;87(19):372-4. No abstract available. German. PMID 4409006